CLINICAL TRIAL: NCT03273140
Title: The Effectiveness of Gamification Diabetes Education Program for Poorly Controlled Type 2 Diabetic Patients: A Randomised Controlled Trial.
Brief Title: The Effectiveness of Gamification Diabetes Education Program for Poorly Controlled Type 2 Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Healthcare Group, Singapore (Other Government)
Collaborators: Tan Tock Seng Hospital (Other)
Responsible Party: Principal Investigator, KHO SIOK EE SHARON, Principal Investigator, Clinical Instructor, National Healthcare Group, Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GDEP
Record Dates: First submitted 2017-08-26; First posted 2017-09-06 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Diabetic Patients, Gamification, Diabetic Education

STUDY DESIGN:
Intervention Model Description: The study adopted a randomized controlled trial (RCT) design, comparing between intervention group (receiving GDEP) and control group (current practice). In this study, the RCT study design allows comparison between the intervention (GDEP), which will then prove the hypotheses and serves to address the aim of this study.
Masking Description: Assessor blinding is not possible as the researcher is involved in the whole process from recruitment to data analysis as part of her doctorate study. However, a research assistant (RA) will assist in arranging the sequence of the envelopes as part of allocation concealment, double-checking of the data entry and analysis of the report. To highlight, the RA will also not know which is the 'control' and 'intervention' group, as both groups will be de-identified as group A and B during the process of data entry and analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gamification Diabetes Education Program (GDEP) (Experimental): The GDEP consists of two components, which are 1) gamification app on diabetes education, and 2) usual care group (face-to-face discussion with a DNE).
  1) Gamification: The development of this gamification app, a mobile-based app of serious gaming, addresses the limitation and few recommendations from the current literature review. It aimed to enhance the user experience, and to facilitate diabetes education in an effective and efficient way, aligning with ADA (2014) guidelines, work instructions, and protocols in one tertiary organization. The learning modules are framed by socio-cognitive framework and self-efficacy. The gaming concept has been implemented into a mobile app, which can be accessed via iOS and Android platforms. It takes an average of 15 minutes to complete per stage. Hence, allowing flexibility for participants to access the games anywhere and anytime using i-pad or mobile devices.
  Interventions: Device: Gamification Diabetes Education Program (GDEP)
- Standard group (No Intervention): The control group comprises of the standard care or usual care group, which is the face-to-face session with the DNE. The content during each session is dependent upon the individual's needs and concerns, including the reason for referral to DNE by the endocrinologist. For example, teaching the individual patient on self-management of blood glucose (SMBG) and emphasizing on diet modification and exercise if necessary. Educational pamphlets on diabetes management will be given to him/her if deemed necessary. Each session will usually requires an average of 45 minutes, which is considered as long consultation that costs 16 dollars. On the other hand, short consultation is categorised as less than 30 minutes that costs around eight dollars. The difference is that there is no GDEP in the control group. However, after the completion of data collection at six months time, the control group will also receive the intervention (GDEP). This is in order to give them equal opportunity.

INTERVENTIONS:
Device: Gamification Diabetes Education Program (GDEP) — "Diabetic application" focuses on diabetes management and consists of two gamelets and consist of story-telling, case scenarios with the integration of problem-based decision-making and solving skills in diabetes management. These scenarios created are familiar to the patients and nurses - to make the games more interactive and realistic to the players (participants). Immediate feedback will be given after they select their decision. The visual reward will appear after attaining one score for each correct question. Participants can easily access and play the games several times till contents are reinforced and knowledge is retained or at their own comfort level. This game mechanics aim to motivate and assist patients to achieve their desired result and self-efficacy behaviors. It addresses the deficits from the current literature review, by aiming to be up-to-date, reliable with new updated scenarios and platform.
  Arms: Gamification Diabetes Education Program (GDEP)

SUMMARY:
Background: The prevalence of DM is increasing across both Asian and Western countries, in proportion to the rising aging population. Type 2 diabetic patients are the high-risk group to experience diabetes-related complications that can lead to depression, poor quality of life and even death. In the current face-to-face diabetes counseling, the patients presented with weak comprehension of diabetes knowledge. There is a gap between application of knowledge and self-efficacy behaviors. With the increased patient acuity in the recent years, it has contributed to the shortage of diabetes nurse educators to meet the demands or needs in the outpatient endocrine clinic. Often, the patients have to wait longer for their turn for diabetes education, which can result in a delay in diabetes self-management. The use of mobile health technologies had demonstrated a positive impact on diabetes-related outcomes and better self-efficacy behaviors, all of which are crucial in diabetes management.

Aims: This study is to evaluate the effectiveness of Gamification Diabetes Education Program (GDEP) on HbA1c values, self-efficacy, sense of coherence and quality of life among the poorly controlled 2 diabetic patients.

Methods: This study adopted a randomized control trial design. Based on Cohen's power analysis, one hundred and forty-eight participants will be recruited through simple random sampling. The recruitment process includes block randomization and allocation concealment. Participants will either be randomized into intervention (GDEP) group or control (current practice) group. The self-efficacy instrument, sense of coherence scale (SOC-13), world health organisation quality of life scale- brief (WHOQoL-BREF) and HbA1c values assessed the outcomes at the same time points: point of enrollment (pre) and two post-time points at 12-week and 24-week.

The significance of study: GDEP would bring about awareness on diabetes management and contribute to existing diabetes literature. It addresses the clinical significance of enhancing diabetes knowledge and motivation in self-efficacy behaviors. Hence, GDEP has the potential to close the gap between application of knowledge to self-efficacy behaviors, which in turn would result in better self-efficacy, sense of coherence and quality of life. All of these could reduce their HbA1c values and the global health care expenditure spent on managing diabetes mellitus alone. The development of GDEP is a value-added and innovative-driven packaging to close the gap and address the limitation in the current literature. It serves to transform workforce and redesign patient education process for type 2 diabetic patients.

DETAILED DESCRIPTION:
The prevalence of Diabetes Mellitus (DM) is increasing internationally, corresponding with the rising aging population. Nearly half of the population was unaware that they have diabetes and the number is portended to reach 439 million worldwide by the year 2030. This global phenomenon draws the attention on the enormous health care expenditure spent on managing DM alone. The financial burden of diagnosed diabetes was 2.3 times higher than the absence of it, reflecting as one of the barriers in engaging diabetes patients and promoting self-efficacy. Type 2 diabetes patients, also known as non-insulin dependent diabetes, are the high-risk population to experience a diabetes-related complication, such as, end-stage renal failure (ESRF), stroke, cardiovascular disease and amputation of the limbs, all of which can lead to poor quality of life (QoL), depression and even death.

Local statistics demonstrated an increase of 25.6% (2013 to 2015) of diabetic patients in an outpatient endocrinology clinic and ten percent hospital readmission rate of patients due to poor compliance and diabetes-related health issues. A retrospective study done locally in the primary health care polyclinics had shown an incline percentage of attendances with DM, from 8.8% to 9.8% over the past five years (2011 to 2015), reflecting an increase of 8155 diabetic patients. Their average age group is 40 years old. According to American Diabetes Association (ADA, 2014), glycosylated hemoglobin A1c (HbA1c) value has been recognized as the standard measurement in diagnosing and treating DM and, the value of ≤7% was correlated with a reduction in diabetes complications. Each 1% of the reduction in HbA1c values over ten years is equivalent to 21% of the reduced risk of diabetes-related outcomes and death, including 14% of the reduced risk for myocardial infarcts and 37% for microvascular complication (p<0.0001). Effective diabetes management or self-efficacy appears strongly related to healthy lifestyle modification and behavioral change, such as medication adherence, compliance to treatment-regime and exercising.

In comparison, poor access to quality care, stress, and obesity has a detrimental effect on HbA1c values and increased the risk for diabetes-related complication as mentioned. Poor clinical outcomes consists of HbA1c >7.0%, systolic blood pressure > 130mmHg, body mass index (BMI) of ≥ 25, abnormal low-density lipoprotein (LDL) and high-density lipoprotein (HDL) measurement. Poor diabetes outcomes are related to depressive symptoms, anxiety, low self-efficacy, poor self-esteem, eating disorders and diabetes-related stress, including osteoporosis among the Chinese diabetes patients. Hence, diabetes patient education is an important cornerstone in self-management, self-efficacy, and long-term behavior change.

Patient education is defined as a process of providing skills and knowledge, including giving advice and alternatives for lifestyle modification in diabetes management and glycemic control. Health education aimed at preventing diabetes-related complications and can lead to improved health literacy that supports greater empowerment in health decision-making and outcomes. There is no consistency of teaching contents in diabetes educational program. It could be due to that the program was led by a different healthcare professional, such as pharmacist, dietician or nutritionist, diabetes nurse educator and or psychologist.

To some extent, the benefits of these diabetes education programs had shown improvement in self-management and glycemic control, including a reduction in depression, and enhancing self-efficacy behaviors and better quality of life. However, all these require an ongoing positive reinforcement in order to achieve a successful long-term intervention and good glycemic control. An effective diabetic patient education would mean success in diabetic self-management, which is associated with better metabolic control, lower costs of therapy through complication prevention, lower mortality rate, reduced readmission rates, improve QoL and, better self-efficacy and health behaviors.

The current diabetic patient education in many hospitals locally, be it private or government sectors still use the traditional teaching method; the face-to-face approach. Primarily and tertiary health care sectors, like polyclinics and outpatient endocrinology clinics, are also using face-to-face approach. There are various health care professionals, such as doctors, nurses, diabetic nurse educator (DNE), dieticians and podiatrists who conduct diabetic education. Face-to-face interactions require intensive manpower, as health care professionals need to engage the patients within a stipulated time period. During these sessions, the DNEs needs to achieve the educational goals, such as impacting knowledge, assessing attitudes and encouraging self-efficacy towards managing their own disease. Each DNE takes an average of 45 minutes in counseling each patient. At times, such educational goals can only be achieved over several scheduled visits, in view of the increasing patient numbers and acuity, and it may not be practical or feasible to achieve the long-term goal with one-time consultation. On the other hand, group based education had demonstrated better health outcomes in HbA1c values, diabetes knowledge, feeling of empowerment and reduced fatigue level although North and Palmer (2015) reported no significant difference (p<0.001) in HbA1c values between individual and group-based diabetes education. Nevertheless, the face-to-face advice remains an important influence on behavioral outcomes through motivation and counseling, and likely to constitute knowledge exchange through diabetes education. This social interaction enhances the quality of life (QoL) and promotes critical reflection upon why and how certain activities occur.

A study conducted in Germany reported that elevated HbA1C value of ≥7% was associated with risk of cognitive-decline and dementia among the diabetes patients. Achieving good HbA1c level can delay the onset of microvascular complication (Venkataraman et al., 2013). Diabetes patient education can improve HbA1C values, be it at the most statistically significant at the third month (p=0.02). The other two studies had also shown a clinical improvement in HbA1C values at the six-month, with a p=0.004 (Jaipakdee et al., 2015) and p<0.05. In comparison, two studies had demonstrated no clinical improvement at the 6-month, with a p= 0.94 and p=0.334 respectively. Similarly, Krebs et al., (2013) had shown insignificant HbA1C values at 9-month (p=0.22) and whereas, Collins-McNeil, Edwards, Batch, Benbow, McDougald, and Sharpe (2012) reported significant result (p=0.1) after a 12-weeks diabetes educational program. There is a positive association (p<0.001) between HbA1C values and motivational factors after adjustment for potential confounders, such as gender, age, body mass index and diabetes knowledge (Nouwen et al., 2011). This means that negative proposition, such as depression, portends poorer control of diabetes mellitus; higher HbA1C values.

The clinical management and advice via the traditional consultation approach are insufficient to achieve good diabetes management and glycemic control (Krebs et al., 2013). There is a gap between applications of knowledge to actualize self-efficacy behaviors among the type 2 diabetic patients. Drawing the voices of diabetes patients' perspective on the barriers to better diabetes management and glycemic control could avoid miscommunication. Most studies had explored the barriers and facilitators in diabetes self-management and education. The facilitators that emerged were having good relationship with health care professionals, simple and practical instructions and favorable community environment, although it was suggested to improve the collaboration between primary and secondary care (Raajimakers et al., 2013). The five barriers that emerged were physical barriers (knowledge deficit), psychological barriers (over dependence on western medication despite disliking them; lack of motivation and self-competency to follow guidelines), social barriers (family role expectations, cuisine culture, lack of trustworthy information sources, confusing health information, lack of awareness of lifestyle programs; prevention initiatives and social support, and communication deficit between patient-practitioner), and care system barriers (restriction of reimbursement regulations). Shen et al. (2013) added that the latter barrier had also resulted in a reduction of filial responsibility in China due to the cultural inferences of the one-child policy. These findings supported that self-efficacy and diabetes knowledge is crucial in diabetes management and control.

The use of smartphones and mobile apps has grown exponentially over the years, with technologies touching the remote corners of the globe. Seidel et al. (2014) echoed that 83% of the high-risk group for type II diabetes (mean age of 52.7 years old) prefers technology-based or telephone-supported program than class-based and that the Asians are more likely to choose technology-based program than the Whites. Apparently, half of the causal gamers (participants) fall within the age range of 35 to 64 years old. Mobile health technologies include telemonitoring, web-based program and mobile platform applications, all of which, had demonstrated a positive impact on diabetes-related outcomes and clinician-related outcomes, by addressing issues related to missing medications and finishing prescribed medication. To elaborate, computer-based technology and web-based program promoted knowledge retention and enhanced diabetes knowledge; behavior and HbA1c level that includes reduced hypoglycemia episodes. Hence, it could be a potential alternative to group lectures for diabetes self-management education.

On the other hand, apps are downloadable programs designed to operate on smartphone operating system, and the use of smartphones apps had sustainable benefits in relation to behavioral change and successfully engage the type 2 diabetics, thereby gaining motivation to interpret and use the contents better accordingly to one's needs. The key point in using mobile apps is to improve user experience so as to enhance engagement. A study conducted in South Caroline reported a 0.5% reduction means of the HbA1c level after mobile health intervention over a six-months follow-up. However, this intervention should not only restrict to sms alone as it offers a new and promising platform for connecting patient to meaningful resources, by serving as a practical bridge between health care and community-based resources that promote diabetic self-efficacy, behavioral modification, and all those related to improving diabetes-related health outcomes. Next, it also has the potential to tailor health communication and transform health service delivery on a global perspective concerns.

Gaming is defined as a tool to present complex and real-world problems, linking theory to real-life situations through the application of principles, theory, and concepts. Gamification involves games that are designed with practical training objective or simulation that includes the presentation of factual knowledge and psychomotor skills. The design of avatars in prototype gamification linked gaming to "real-life" situations or clinical settings, and thus, allowing for a more realistic interface to the players. Their advantages are in enhancing the learners' skills through mastery performance, and comprehension of diabetes-related knowledge through observational learning at own pace.

Games may be served as an assessment tool and are good resources for people with lower literacy level as it permits repetitive usage and learning at own pace. The more the participants engaged with games, the higher the sense of being "in control", "important" and "empowered". In contrast, the longer the duration of attention retention through games, the greater the exposure and likelihood of a behavior change. The effectiveness of gaming was reflected by an improvement seen in self-efficacy, symptom management and knowledge gained through active participation. Games can also address few unmet needs, such as, retaining of contents and information through repetitive playing and learning; compare and contrast information resource; allowing clinicians to keep tracks on the games scores; a sense of control over own body and challenging reality of everyday life.

Another important key aspect to take note when developing informatics technology, is the health status of an individual, in view that the diabetes people with disabilities are less likely to use the internet than others due to the lack of access, expertise and physical conditions that made the Internet use difficult. There was a study limitation in reporting the effectiveness and feasibility of games for type 2 diabetes patients. Eagleson et al. (2017) supported that the development and implementation of mobile health and web-based interventions are not well documented and fragment in the current literature. The concerns being raised were that either the mobile application was developed in an American context with different guideline recommendations that may influence the effectiveness and utility in different context, or that, the gaming platforms were either outdated or short shelf life, which can result in confusion due to uncertainty about reliability, security, regulation and integration concerns. In addition, the games are also not updated with new scenarios regularly on a long-term basis.

The other flip sides of mobile gaming application include the inability to address the psychological (human factors), motivation, provider-patient miscommunication (health care system) and social-economic aspects, which can affect self-management or manageability, and that, it can be costly and time-consuming in the development process. It was recommended to consider these prior developing a gaming application, which were (i) using a highly personalized and user-centered system for compliance and educational needs, (ii) input an interactive tool, such as dragging food into a plate, (iii) input a nursing workstation for accessibility of information and problem-solving solutions, and lastly, (iv) input sharing forum and interactive quizzes.

Mobile apps could be an innovative way of learning or packaging in diabetes education. Although a pilot study conducted in California reported that their bilingual diabetic program demonstrated that improved knowledge might not be required to improve positive behaviors, but it aids in preventing errors while using diabetes technology. Individual using technology has a better understanding and knowledge on DM. The impact of increased knowledge can firstly, influence the individual's understanding and perception of how diabetes is being viewed, based on one's experience and the information retrieved from social media, family and friends, especially those with diabetes. This, in turn, can either act as a motivator or barrier to their cognitive domain. The challenge ahead is to implement steps to trigger the meaningfulness out from that individual, so as to engage him/her in lifestyle modification and taking ownership of own health, such as healthy eating, foot care, and medication adherence. Secondly, knowledge influence individual's adherence to medication, self-care and treatment plan, which can enhance HbA1C level, and promote self-efficacy and health behaviors, such as self-monitoring of blood glucose level. Diabetes patients feel empowered once they have sufficient knowledge to make rational decisions, sufficient control, and resources to implement their decisions, and sufficient experience to evaluate the effectiveness of their decision. Thus, enhance QoL and reduces mental health concerns, such as anxiety and depression. Improving the quality of life could result in better motivation and social activity.

There is a dearth of knowledge on in these areas: firstly, there is a study limitation in integrating socio-cognitive framework and self-efficacy into designing a gamification diabetic educational program, which includes evaluating its feasibility as an assessment tool in diabetes education. Secondly, there is a lack of uniformity and consistency in teaching contents, delivery of health policy and culturally congruent services in a multi-facet country. Thirdly, there is a study limitation in using randomized control trial design to evaluate the effectiveness of the empirical gamification diabetes educational program on HbA1c values, self-efficacy, sense of coherence and quality of life. This study will firstly, add to the growing research on using gamification application as an education tool in the diabetic population, and secondly, serves to transform workforce and redesign patient education process for type II diabetes patients that include achieving optimum productivity and delivering of value-added services that meet the needs of the future healthcare system.

ELIGIBILITY:
Inclusion Criteria:

1. Patient who is clinically diagnosed with type 2 diabetes mellitus.
2. Patient with HbA1C value > 7% at least within the past two months.
3. Patient who can speak and understand English.
4. Patient of age 21 to 75 years old.
5. Patient with either a smartphone or i-pad/ tablet.

Exclusion Criteria:

1. Pregnant patient.
2. Patient diagnosed to have a terminal illness.
3. Patient with cognitive impairment.
4. Patient with end-stage renal failure (ESRF).

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2018-08-15 (Actual)

PRIMARY OUTCOMES:
Better HbA1c values | Every three months up to 24th week (0 week as baseline, 12th week and 24th week)
  Clinical indicator to monitor glycemic control for the past three months
Better Self-efficacy | Every three months up to 24th week (0 week as baseline, 12th week and 24th week)
  Using Self-efficacy tool (Duprez et al., 2013)
Better Sense of Coherence | Every three months up to 24th week (0 week as baseline, 12th week and 24th week)
  Using SOC-13

SECONDARY OUTCOMES:
Better Quality of life | Every three months up to 24th week (0 week as baseline, 12th week and 24th week)
  Using genetic tool: WHO-BREF

CONTACTS AND LOCATIONS:
Locations (1):
- 11 Jalan, Tan Tock Seng Hospital,, Singapore, Noverna, Singapore

IPD SHARING:
Plan to Share IPD: No